CLINICAL TRIAL: NCT02768324
Title: the Effect of Gut Microbiota on the Prognosis of Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jinan University Guangzhou (Other)
Responsible Party: Principal Investigator, Deng Li, Ph.D. student, Jinan University Guangzhou
Other Study IDs: 13123412341
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Sepsis
Keywords: sepsis; Gastrointestinal Microbiome; Gut microbiota; Gut Flora; Intestinal Flora
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- sepsis with diarrhea
- sepsis without diarrhea

SUMMARY:
Sepsis is a life-threatening condition that arises when the body's response to infection injures its own tissues and organs. Common signs and symptoms include fever, increased heart rate, increased breathing rate, and confusion. Clinically, sepsis patients with diarrhea often result in a bad prognosis. Gut microbiota consists of a complex community of microorganisms that live in the digestive tracts of animals. The gut microbiota comprises the largest and most diverse reservoir of mutualistic microorganisms associated with animals. The aims of this study is to determin the effect of gut microbiota on the prognosis of Sepsis, by using 16s pyrosequencing, comparing the blood culture result.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with sepsis
* 18 years to 65 years of age

Exclusion Criteria:

* patients had complications such as acute cerebral infarction or acute myocardial infarction
* The use of antibiotics, pro-prebiotics within 3 months
* <18 years or >65 years
* History of intestinal surgery
* patients withdraw from this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with sepsis were included in this study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Discharged from ICU | 7 days